CLINICAL TRIAL: NCT04816383
Title: A Smartphone-Based Approach to Improved Breast-Feeding Rates And Self-Efficacy: A Randomized Controlled Clinical Trial
Brief Title: A Smartphone-Based Approach to Improved Breast-Feeding Rates And Self-Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Carolyn Zahler-Miller, Assistant Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1699671
Record Dates: First submitted 2021-03-20; First posted 2021-03-25 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Breastfeeding
Keywords: smartphone application; breastfeeding; breastfeeding self-efficacy
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Control group will usual breastfeeding care (counseling by provider, access to lactation consultant, etc) Interventional group will receive usual care plus the breastfeeding application introduced between 32 to 36 weeks estimated gestational age.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The participant cannot be blinded as they will be using the application. The investigator cannot be blinded as they have to provide the application to the patient, teach them how to use it, and perform their surveys about the application use.
  The outcomes assessor and care provider will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): The participant will receive usual breastfeeding care such as counseling by her physician, access to lactation consults, nursing assistance in the hospital, access to our online resources. The participant will also receive the Apple breastfeeding application in the office once enrolled in the study between 32 to 36 weeks gestation. The participant will be taught how to use the application, and will have access to the study to continue use throughout the duration of follow-up.
  Interventions: Other: "Breastfeeding at AU" Apple-Based Smartphone Application
- Control Arm (No Intervention): The participant will receive usual breastfeeding care such as counseling by her physician, access to lactation consults, nursing assistance in the hospital, access to our online resources.

INTERVENTIONS:
Other: "Breastfeeding at AU" Apple-Based Smartphone Application — This is a free Apple-Based Smartphone Application the participant can download. In the application, there is information and tips for breastfeeding success and continuation, as well as information on additional resources both online and in the community as a whole.
  Arms: Experimental Arm

SUMMARY:
To provide patients with easily accessible information in the form of a smartphone application regarding medically appropriate information about breastfeeding and to assess the impact this information has on women's breastfeeding rates and perception of self-efficacy.

DETAILED DESCRIPTION:
The benefits of breastfeeding for both mother and neonate have been well documented and extensively researched. Breastfeeding rates remain suboptimal despite known advantages including reduced lifetime risk of maternal ovarian cancer, more rapid return to pre-gestational weight, improvement in maternal/neonatal bonding, reduction in neonatal allergic/immunologic conditions. Both non-modifiable and modifiable factors affecting a mother's decision regarding breastfeeding have been identified. Modifiable factors include breastfeeding knowledge, self-efficacy, and confidence. Breastfeeding self-efficacy has been positively correlated with breastfeeding duration. There is a lack of local data on breastfeeding rates, duration, and self-efficacy in the Augusta University women's health population as well as a lack of documented improvement of these factors following educational programs. Our study aims to create a program that is easily accessible and available to our patient population in the form of a free application available on Apple devices capable of accessing the internet (e.g., i-phone, i-pad, etc.). This study will be a randomized control trial. The intervention group will have access to the application while the control group will not. Our hypothesis is that the application will improve long-term breastfeeding rates, duration, and self-efficacy if offered to patients at 32 through 36 weeks gestation. This will be assessed by comparing initial self-efficacy survey results with survey results at 12 months postpartum for the intervention versus control groups. We will also measure breastfeeding duration during the first 12 months postpartum and exclusive breastfeeding rates at 6 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous and multiparous females receiving prenatal care at Augusta University Obstetrics and Gynecology clinic at 32 through 36 weeks gestation.
* No documented anatomic differences in mother's chest anatomy.
* Access to the internet via an Apple® device (such as i-phone or i-pad).
* Delivery at Augusta University Medical Center

Exclusion Criteria:

* Significant maternal intrapartum or postpartum complications (i.e., postpartum hemorrhage > 2000 mL, uterine inversion, retained products, ICU admission, postpartum psychosis).
* Infants admitted to neonatal intensive care unit >48 hours
* Pre-term deliveries prior to 37 weeks gestation
* Infants with cleft palate, or other palate/facial defects
* Patients without email access or internet access
* Patients without an Apple® device (i-phone, i-pad)
* Non-English speaker
* Mothers unable to breastfeed secondary to contraindicated communicable disease (i.e.

HIV)

* Mothers unable to breastfeed secondary to contraindicated medications
* Mothers of infants up for adoption

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — This project is aimed at postpartum women and the application's effect on breastfeeding rates.
Enrollment: 93 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Breastfeeding duration | 12 months postpartum
  We will assess total breastfeeding duration

SECONDARY OUTCOMES:
Breastfeeding Self-Efficacy Rates | 12 months postpartum
  The breastfeeding self-efficacy short form is a validated, standardized form to assess participants' sense of breastfeeding self-efficacy.

OTHER OUTCOMES:
Breastfeeding Rates | 6 months postpartum
  We will assess the exclusive breastfeeding rates at 6 months postpartum
Breastfeeding Rates | 12 months postpartum
  We will assess the exclusive breastfeeding rates at 12 months postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Mello Sa SR, Wang Z, Sapkalova V, Sullivan M, Saucedo Baza A, Delgado P, Looney S, Zahler-Miller C. A smartphone-based application to improve breastfeeding duration and self-efficacy: a randomized controlled clinical trial. Women Health. 2025 Feb;65(2):154-166. doi: 10.1080/03630242.2024.2448519. Epub 2025 Jan 3. PMID 39748676